CLINICAL TRIAL: NCT04833036
Title: Second-line Irinotecan Combined With Cetuximab (c-CetuIRI) Versus Second-line Irinotecan Three-line Irinotecan Plus Cetuximab (s-IRI-CetuIRI) in the Treatment of Oxaliplatin and 5-FU Phase II Clinical Study of Wild-type Advanced Colorectal Cancer With RAS Gene
Brief Title: c-CetuIRI Versus Ersecond-line Irinotecan s-IRI-CetuIRI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cetu-IRI
Record Dates: First submitted 2019-10-12; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer
Keywords: chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- c-CetuIRI (Active Comparator): Irinotecan combined with cetuximab
  Interventions: Drug: Irinotecan; Drug: cetuximab
- s-IRI-CetuIRI (Experimental): single irinotecan first, then irinotecan plus cetuximab sequentially after PD
  Interventions: Drug: Irinotecan; Drug: cetuximab

INTERVENTIONS:
Drug: Irinotecan — 180 mg/m2, ivgtt d1，q2w
Drug: cetuximab — 500 mg/m2, ivgtt d1，q2w

SUMMARY:
The primary endpoint is to evaluate the progression-free survival (PFS).

DETAILED DESCRIPTION:
This study was designed for patients with advanced bowel cancer after first-line LOHP and 5-FU treatment failure. The control group was treated with second-line CPT-11+C225. The study group used second-line CPT-11 single drug until the third line was CPT-11+C225. treatment. Referring to the previous literature data, the PFS of the second-line treatment of CPT-11+C225 is about 4 months. This study assumes that the total PFS time of C225 can be extended to 7 months after the failure of second-line CPT-11 treatment compared with the direct second-line combination. , set α = 0.05, β = 0.2, the expected enrollment time is 2 years, the follow-up time is 1 year, the 10% sample shedding rate, the total sample size is about 60 cases per group, a total of 120 cases.

ELIGIBILITY:
Inclusion Criteria:

1. Signing informed consent;
2. Age is greater than or equal to 18 years old;
3. Metastatic colorectal adenocarcinoma confirmed by tissue or cytopathology;
4. First-line failure to use oxaliplatin combined with fluorouracil (with or without anti-angiogenic targeting drugs);
5. One or more measurable lesions, the longest diameter of the spiral CT scan is at least 10 mm, and the diameter of the conventional CT scan is at least 20 mm (the solid tumor efficacy evaluation standard, RECIST standard, version 1.1);
6. The Eastern Cancer Cooperative Group (ECOG) has a general status score of 0-2;
7. The bone marrow capacity, liver and kidney function reached the following criteria within 7 days before screening:

   Absolute neutrophil count ≥ 1.5x109 / L; hemoglobin ≥ 9.0 g / dl; platelet count ≥ 80 x 109 / L; total bilirubin ≤ 1.5 times normal upper limit (ULN); alanine aminotransferase and aspartate aminotransferase ≤ 2.5 x ULN Alkaline phosphatase ≤ 3 x ULN; serum creatinine ≤ 1.5 x ULN;
8. Women of childbearing age need to take effective contraception.
9. RAS, B-RAF gene wild type

Exclusion Criteria:

1. Previous use of irinotecan or anti-egfr therapy for advanced colorectal cancer (e.g. Cetuximab, panizumab, etc.);
2. History of HIV infection or active chronic hepatitis b or c (high copy viral DNA);
3. Patients with important organ failure or other important diseases: patients with serious heart disease including congestive heart failure, uncontrolled arrhythmia, angina requiring long-term medication, heart valve disease, myocardial infarction, pericardial effusion with obvious symptoms, and refractory hypertension;A history of severe neurological or psychiatric problems;Severe infection;Active disseminated intravascular coagulation
4. Active severe clinical infection;
5. Symptomatic brain or meningeal metastasis (unless the patient was treated for > for 6 months, had negative imaging results within 4 weeks prior to study entry, and had stable tumour-related clinical symptoms at study entry);
6. Patients whose seizures require treatment (e.g. steroids or antiepileptic therapy);
7. Receiving renal dialysis;
8. Have a history of other malignant tumors within 5 years, except for cured cervical carcinoma in situ or skin basal cell carcinoma, except for those whose metastasis can be confirmed by pathology to be from other tumor sources;
9. Chronic intestinal diseases, infectious intestinal diseases and intestinal obstruction;
10. Drug abuse and medical, psychological or social conditions may interfere with patients' participation in studies or affect the assessment of their findings;
11. Any unstable condition or condition that may endanger the safety and compliance of patients;
12. Pregnant or lactating women;Having fertility but not taking adequate contraceptive measures;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 8 weeks
  progression free survival

SECONDARY OUTCOMES:
OS | through study completion, an average of half year
  overall survival
ORR | up to 8 weeks
  objective response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China